CLINICAL TRIAL: NCT06192329
Title: Hot Water Therapy for the Treatment of Menopause-related Hot Flashes and Other Symptoms: a Clinical Trial
Brief Title: Hot Water Therapy for the Treatment of Menopause-related Hot Flashes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Colorado Springs (Other)
Collaborators: East Carolina University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-029-HYBL
Record Dates: First submitted 2023-12-01; First posted 2024-01-05 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Menopause; Menopause Related Conditions; Menopause Syndrome
Keywords: heat therapy; hot water therapy; hot water immersion; vasomotor syndrome; hot flashes; hot flushes
MeSH Terms: conditions — Hyperthermia; Hot Flashes | interventions — Diathermy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Warm water immersion (Sham Comparator): On days 2-6 and 8-12 of the therapy sessions, the participants will immerse themselves up to the shoulder in 97°F water for ~30 min, followed by immersion to the hip level for ~60 min (total immersion time of 90 min).
  Interventions: Behavioral: Warm water immersion
- Hot water immersion (Experimental): On days 2-6 and 8-12 of the therapy sessions, the participants will immerse themselves up to the shoulder in 105°F water for ~30 min, followed by immersion to the hip level for ~60 min (total immersion time of 90 min).
  Interventions: Behavioral: Hot water therapy

INTERVENTIONS:
Behavioral: Hot water therapy — On days 2-6 and 8-12 of the therapy sessions, the participants will immerse themselves up to the shoulder in 105°F water for ~30 min, followed by immersion to the hip level for ~60 min (total immersion time of 90 min).
  Other Names: heat therapy; hot water immersion
  Arms: Hot water immersion
Behavioral: Warm water immersion — On days 2-6 and 8-12 of the therapy sessions, the participants will immerse themselves up to the shoulder in 97°F water for ~30 min, followed by immersion to the hip level for ~60 min (total immersion time of 90 min).
  Other Names: Control trial; Sham trial
  Arms: Warm water immersion

SUMMARY:
The purpose of this research is to determine whether hot water therapy (i.e. taking prolonged hot baths on multiple consecutive days) decreases hot flash symptoms and improves mood in women who are undergoing or who have underwent menopause. It is hypothesized that women who undergo hot water therapy will have reduced hot flash symptoms and improved mood.

Initial tracking period: Women who volunteer to participate in this study will be asked to track the frequency and intensity of their hot flash and other menopause-related symptoms for an initial two week period. Afterwards, they will start their heat therapy program.

Physiological assessments: On days 1, 7, and 13 of the heat therapy sessions, the participants will enter a climate controlled room to have their thermoregulatory responses assessed. This will consist of slowly walking on a motorized treadmill in 99.5°F (37.5°C) and 30% relative humidity conditions, for 30 min, after which the humidity in the climate chamber will be progressively increased until their core temperature begins to increase (~2 hour total time). Before and/or during these trials, core temperature, heart rate, whole-body sweat losses, thermal comfort, local sweat rate, and skin blood flow will be measured, and a 6 ml (~1 tsp) blood sample will be taken, to assess how the participants respond to the heat stress. These sessions should take less than 3 hours to complete.

Hot water therapy sessions: Upon enrolling in the study, the participants will be assigned to one of two groups: water bathing at 105°F or 97°F in the lab. On days 2-6 and 8-12 of the therapy sessions, the participants will immerse themselves to a water level at the shoulders for ~30 min, followed by immersion to the hip level for ~60 min (total immersion time of 90 min).

Post-intervention tracking period: after completing the heat therapy sessions, the participants will be asked to continue to take baths at home once every 4 days for 1 month. During this time, the participants will be asked to record the intensity and frequency of their hot flashes daily and other menopause-related symptoms weekly. At the end of this month the participants will be given a final exit survey, in order for them to provide the researchers information about their experience participating in the study.

DETAILED DESCRIPTION:
Menopause is the time at which menstruation stops and perimenopause is the period before, characterized by a continuous reduction in estrogen and progesterone levels in the blood. Concurrently, the reductions in estrogen leads to a rise in another hormone, orexin. The reduction in circulating estrogen and progesterone and the increase in circulating orexin have been demonstrated to play a major role in menopause-related hot flashes and night sweats, known as vasomotor symptoms (VMS), as well as other symptoms such as mood disorders.

While hormonal replacement therapy remains the most effective defense against VMS, there has been a progressive decline in its prescription due to side effects such as uterine bleeding, increased risk of thromboembolism, as well as increased rates of gallbladder, breast, endometrial, and urinary cancers, highlighting the need for alternative non-hormonal treatments.

Exercise, and specifically the thermoregulatory benefits of exercise (i.e. increased sweating and skin blood flow, as well as reduced core temperature), improves vasomotor symptoms in women going through menopause. Heat acclimation/heat therapy improves thermoregulatory responses by more than twice as much as exercise alone, however, to date, no studies have investigated the effects of heat acclimation on menopause-related vasomotor symptomology.

Accordingly, the purpose of this study will be to examine whether hot water bathing improves vasomotor symptomology, with the guiding hypothesis that hot water bathing will reduce vasomotor symptomology.

Recruitment For this study, we will aim to recruit 100 women who have either undergone or who are undergoing menopause and who self-report experiencing vasomotor symptomology.

Study protocol An initial visit will be organized during which the potential participants will complete a health screening and consent to participate in the study. After which, the participants will undergo a two week-long baseline period during which they will track their vasomotor symptomology using a vasomotor symptomology journaling template, as well as complete a standardized menopause symptomology questionnaire. The participants will be randomized into two groups: a hot water bathing group and a sham group.

Following the baseline period, participants will report to the climate chamber located in the Hybl center to have their thermoregulatory responses assessed. This will consist of slowly walking on a motorized treadmill in 99.5°F (37.5°C) and 30% relative humidity conditions, for 30 min after which the humidity in the climate chamber will be progressively increased until an inflection in the participants' core temperature is detected. Before and/or during these trials, core temperature, heart rate, whole-body sweat losses, thermal comfort, local sweat rate, and skin blood flow will be measured, and a 6 ml (~1 tsp) blood sample will be taken, to assess heat loss adaptations.

Next, the participants will begin their 10-day, hot water bathing sessions. The participants in the treatment group will be asked to submerge themselves in a bathtub filled with 105°F (40.5°C) water, and to remain at this depth until their esophageal temperature reaches 101.5°F (38.6°C). Based on previous hot water therapy studies using this protocol, this should take approximately 25-35 min. After attaining the target core temperature, the participants will be given a stool to sit on in order for them to remain at waist depth in the water in order to maintain their core temperature at 101.5°F (38.6°C) for an additional 60 min. Participants in the sham group will be immersed up to the shoulder in a 97°F (36°C) tub for 30 min and then to waist-level for another 60 min in order to mimic the same hydrostatic pressures as were experienced by the participants in the heat therapy group, but without the heat exposure.

Finally, following the heat therapy sessions, the participants will be asked to take hot baths at home once every four days (as this is the frequency needed to stay heat acclimated) for one month, while continuing to track their vasomotor symptomology. At the completion of this follow up period, they will complete a study exit survey that has questions regarding their experience in the study.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported menopause-related hot flashes

Exclusion Criteria:

* Diagnosed with a cardiovascular illness that precludes them from taking part in exercise

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Greene climacteric questionnaire | One month pre therapy through to one month post therapy
  This is a standard questionnaire used to quantify the intensity of 21 common menopause-related symptoms. The score for each question ranges in intensity from 0 (not at all) to 3 (extremely).
Daily hot flash diary | One month pre therapy through to one month post therapy
  Based on industry-standard hot flash diaries, this tracks the number and intensity (where 1 is none and 10 is extreme) of hot flashes, night sweats, and mood disruptions that the participants feel.

SECONDARY OUTCOMES:
Core temperature | Day zero, six, and 12 of therapy
  Measured using esophageal and rectal probes. Indicator of physiological heat acclimation status.
Maximum skin wettedness | Day zero, six, and 12 of therapy
  Maximum skin wettedness is a measure of how much of a person's skin surface they are able to wet through sweating. In an inactive, non-heat acclimated person, a normal skin wettedness value is approximately 70%. In an active, fully-heat acclimated person, a normal skin wettedness value is approximately 100%. Skin wettedness is determined by having a person walk at a constant speed on a treadmill in a 37.5degC climate chamber, while humidity levels are progressively increased. Maximum skin wettedness is determined from the humidity level in the climate chamber at which the participant's core temperature begins to rise. The more heat acclimated a person is, the higher the humidity will get to in the room before their core temperature rises.
Blood plasma volume | Day zero, six, and 12 of therapy
  Determined from venous blood draws. Indicator of physiological heat acclimation status.
Sweat rate | Day zero, six, and 12 of therapy
  Both whole-body using a high-precision platform scale and locally using the ventilated capsule technic. Indicator of physiological heat acclimation status.
Skin blood flow | Day zero, six, and 12 of therapy
  Determined using laser doppler flowmetry. Indicator of physiological heat acclimation status.
Reproductive hormone levels (estrogen, progesterone, luteinizing hormone, orexin) | Day zero, six, and 12 of therapy
  Determined from venous blood draws. Indicator hormonal status

OTHER OUTCOMES:
Exit questionnaire | One month post therapy
  Further questions for the participants to complete once at the end of the study in order to gain insight into their subjective experiences using heat therapy and to determine the likelihood the participants would implement this therapy in their lives.

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Morris, PhD, Principal Investigator — University of Colorado, Colorado Springs
Locations (1):
- Hybl Sports Medicine and Performance Center, Colorado Springs, Colorado, United States

DOCUMENTS (1):
  • Informed Consent Form (2023-09-21): https://cdn.clinicaltrials.gov/large-docs/29/NCT06192329/ICF_000.pdf